CLINICAL TRIAL: NCT02211209
Title: A Randomized, Double-Blind, Placebo-Controlled, Phase 3 Study of ISIS 304801 Administered Subcutaneously to Patients With Familial Chylomicronemia Syndrome (FCS)
Brief Title: The APPROACH Study: A Study of Volanesorsen (Formerly IONIS-APOCIIIRx) in Patients With Familial Chylomicronemia Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ionis Pharmaceuticals, Inc. (Industry)
Collaborators: Akcea Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ISIS 304801-CS6; 2014-002421-35 (EudraCT Number)
Record Dates: First submitted 2014-08-05; First posted 2014-08-07 (Estimated); Results first posted 2022-04-13 (Actual); Last update posted 2022-04-13 (Actual); Status verified 2022-03

CONDITIONS: Familial Chylomicronemia Syndrome
MeSH Terms: conditions — Familial hyperchylomicronemia syndrome | interventions — ISIS 304801; Apolipoprotein C-III

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Volanesorsen-matching placebo administered subcutaneously once-weekly for 52 weeks.
  Interventions: Drug: Placebo
- Volanesorsen (Experimental): Volanesorsen 300 mg administered subcutaneously once-weekly for 52 weeks.
  Interventions: Drug: Volanesorsen

INTERVENTIONS:
Drug: Volanesorsen
  Other Names: ISIS 304801; ApoC-III; Approach; IONIS-APOCIIIRx
  Arms: Volanesorsen
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of volanesorsen given for 52 weeks in participants with Familial Chylomicronemia Syndrome

ELIGIBILITY:
Inclusion Criteria:

* History of chylomicronemia
* A diagnosis of Familial Chylomicronemia Syndrome (Type 1 Hyperlipoproteinemia)
* Fasting triglycerides (TG) ≥ 750 mg/dL (8.4 mmol/L) at Screening

Exclusion Criteria:

* Diabetes mellitus if newly diagnosed or if HbA1c ≥ 9.0%
* Other types of severe hypertriglyceridemia
* Active pancreatitis within 4 weeks of screening
* Acute Coronary Syndrome within 6 months of screening
* Major surgery within 3 months of screening
* Treatment with Glybera therapy within 2 years of screening
* Previous treatment with IONIS-APOCIIIRx
* Have any other conditions in the opinion of the investigator which could interfere with the participant participating in or completing the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2016-12-19 (Actual); Study Completion 2017-03-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (38):
- United States (11):
  - IONIS Investigative Site, Encinitas, California
  - IONIS Investigative Site, San Francisco, California
  - IONIS Investigative Site, Kansas City, Kansas
  - IONIS Investigative Site, Boston, Massachusetts
  - IONIS Investigative Site, New York, New York
  - IONIS Investigative Site, Oklahoma City, Oklahoma
  - IONIS Investigative Site, Portland, Oregon
  - IONIS Investigative Site, Philadelphia, Pennsylvania
  - IONIS Investigative Site, Houston, Texas
  - IONIS Investigative Site, Norfolk, Virginia
  - IONIS Investigative Site, Seattle, Washington
- Brazil (2):
  - IONIS Investigative Site, Campinas
  - IONIS Investigative Site, São Paulo
- Canada (3):
  - IONIS Investigative Site, Vancouver, British Columbia
  - IONIS Investigative Site, Chicoutimi, Quebec
  - IONIS Investigative Site, Sainte-Foy, Quebec
- France (3):
  - IONIS Investigative Site, Marseille
  - IONIS Investigative Site, Nantes
  - IONIS Investigative Site, Paris
- Germany (2):
  - IONIS Investigative Site, Berlin
  - IONIS Investigative Site, Dresden
- IONIS Investigative Site, Szikszó, Hungary
- IONIS Investigative Site, Safed, Israel
- Italy (3):
  - IONIS Investigative Site, Milan
  - IONIS Investigative Site, Palermo
  - IONIS Investigative Site, Rome
- Netherlands (2):
  - IONIS Investigative Site, Amsterdam
  - IONIS Investigative Site, Rotterdam
- IONIS Investigative Site, Cape Town, South Africa
- Spain (6):
  - IONIS Investigative Site, Zaragoza, Aragon
  - IONIS Investigative Site, A Coruña, Galicia
  - IONIS Investigative Site, Barcelona
  - IONIS Investigative Site, Madrid
  - IONIS Investigative Site, Málaga
  - IONIS Investigative Site, Seville
- United Kingdom (3):
  - IONIS Investigative Site, Birmingham
  - IONIS Investigative Site, Manchester
  - IONIS Investigative Site, Peterborough

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Witztum JL, Gaudet D, Freedman SD, Alexander VJ, Digenio A, Williams KR, Yang Q, Hughes SG, Geary RS, Arca M, Stroes ESG, Bergeron J, Soran H, Civeira F, Hemphill L, Tsimikas S, Blom DJ, O'Dea L, Bruckert E. Volanesorsen and Triglyceride Levels in Familial Chylomicronemia Syndrome. N Engl J Med. 2019 Aug 8;381(6):531-542. doi: 10.1056/NEJMoa1715944. PMID 31390500
- [Derived] Prohaska TA, Alexander VJ, Karwatowska-Prokopczuk E, Tami J, Xia S, Witztum JL, Tsimikas S. APOC3 inhibition with volanesorsen reduces hepatic steatosis in patients with severe hypertriglyceridemia. J Clin Lipidol. 2023 May-Jun;17(3):406-411. doi: 10.1016/j.jacl.2023.04.007. Epub 2023 Apr 27. PMID 37164837
- [Derived] Hegele RA, Berberich AJ, Ban MR, Wang J, Digenio A, Alexander VJ, D'Erasmo L, Arca M, Jones A, Bruckert E, Stroes ES, Bergeron J, Civeira F, Witztum JL, Gaudet D. Clinical and biochemical features of different molecular etiologies of familial chylomicronemia. J Clin Lipidol. 2018 Jul-Aug;12(4):920-927.e4. doi: 10.1016/j.jacl.2018.03.093. Epub 2018 Apr 4. PMID 29748148
- [Derived] Digenio A, Dunbar RL, Alexander VJ, Hompesch M, Morrow L, Lee RG, Graham MJ, Hughes SG, Yu R, Singleton W, Baker BF, Bhanot S, Crooke RM. Antisense-Mediated Lowering of Plasma Apolipoprotein C-III by Volanesorsen Improves Dyslipidemia and Insulin Sensitivity in Type 2 Diabetes. Diabetes Care. 2016 Aug;39(8):1408-15. doi: 10.2337/dc16-0126. Epub 2016 Jun 6. PMID 27271183

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 67 participants were randomized at 40 study centers in the United States, Canada, Brazil, France, Germany, Israel, Italy, Netherlands, South Africa, Spain, and the United Kingdom.
Pre-assignment Details: 67 participants were randomized, and 66 received study drug. The study included an 8-week screening period (including a diet-stabilization period), a 52-week treatment period, and a 13-week post-treatment evaluation period.
Period: Overall Study
Arm/Group | Placebo | Volanesorsen
Started | 34 | 33
Dosed | 33 | 33
Completed | 32 | 19
Not Completed | 2 | 14
Not completed — Investigator judgment | 0 | 1
Not completed — Voluntary withdrawal | 1 | 4
Not completed — Adverse Event or Serious Adverse Event | 0 | 9
Not completed — Reason Not Specified | 1 | 0

BASELINE CHARACTERISTICS:
Population: The safety set included all randomized participants who received at least one dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Volanesorsen | Total
Number analyzed (Participants) | 33 | 33 | 66
Age, Continuous [Mean (Standard Deviation); unit: years] | 46 (14) | 47 (13) | 46 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 17 | 36
  Male | 14 | 16 | 30
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 7 | 14
  Not Hispanic or Latino | 26 | 26 | 52
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 29 | 24 | 53
  Asian | 4 | 7 | 11
  Other Race | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  Canada | 8 | 6 | 14
  Netherlands | 1 | 3 | 4
  United States | 6 | 5 | 11
  Brazil | 0 | 2 | 2
  Italy | 5 | 5 | 10
  United Kingdom | 3 | 5 | 8
  South Africa | 1 | 1 | 2
  Israel | 0 | 1 | 1
  France | 3 | 3 | 6
  Germany | 0 | 1 | 1
  Spain | 6 | 1 | 7
Fasting Triglycerides [Mean (Standard Deviation); unit: milligrams per deciliter (mg/dL)] | 2152 (1153) | 2267 (1259) | 2209 (1199)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Fasting Triglycerides (TG) From Baseline to Month 3
Description: The Month 3 endpoint was defined as the average of Week 12 (Day 78) and Week 13 (Day 85) fasting assessments.
Time Frame: Baseline to 3 months
Population: The full analysis set included all participants who were randomized, received at least one dose of study drug, and had a baseline TG assessment.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Placebo | Volanesorsen
Number analyzed (Participants) | 33 | 33
percent change | 17.6 [-4.0 to 39.2] | -76.5 [-97.4 to -55.5]
Statistical Analysis 1: Comparison: Placebo vs Volanesorsen; Test type: Superiority; p < 0.0001, ANCOVA; Least Squares Mean Difference = -94.1, 95% CI 2-sided [-121.7 to -66.6]

2. Secondary Outcome: Change From Baseline in Postprandial TG Area Under the Curve (AUC)(0-9h)
Description: Participants had 2 postprandial assessments - one at Baseline (completed at least 48 hours prior to first dose) and one at any time between Week 13 and 19, inclusive. Assessment timepoints include from 1-hr before to up to 9 hrs after ingestion of the meal at 1-hour interval. Postprandial AUC results were calculated using a linear trapezoidal rule for each postprandial measure in the subset of participants who had postprandial assessments 0-9 hour results at baseline and the postbaseline between Week 13 to 19.
Time Frame: Baseline to an on-treatment assessment between Week 13 and Week 19
Population: The full analysis set included all participants who were randomized, received at least one dose of study drug, and had a baseline TG assessment. Data were reported for evaluable participants.
Measure: Mean (Standard Deviation); unit: millimole hours per liter (mmol*h/L)
Arm/Group | Placebo | Volanesorsen
Number analyzed (Participants) | 11 | 10
millimole hours per liter (mmol*h/L) | 36.92 (121.54) | -234.77 (94.86)

3. Secondary Outcome: Absolute Change From Baseline in Fasting TG at Month 3
Description: The Month 3 endpoint was defined as the average of Week 12 (Day 78) and Week 13 (Day 85) fasting assessments.
Time Frame: Baseline to 3 months
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Placebo | Volanesorsen
Number analyzed (Participants) | 33 | 33
mg/dL | 92 [-301 to 486] | -1712 [-2094 to -1330]
Statistical Analysis 1: Comparison: Placebo vs Volanesorsen; Test type: Superiority; p < 0.0001, ANCOVA; Least Squares Mean Difference = -1804, 95% CI 2-sided [-2306 to -1302], Standard Error of Mean 251

4. Secondary Outcome: Treatment Response Rate Defined as Participants With Fasting Plasma TG < 750 mg/dL at Month 3
Description: The Month 3 endpoint was defined as the average of Week 12 (Day 78) and Week 13 (Day 85) fasting assessments. mg/dL = milligrams per deciliter
Time Frame: Baseline to 3 months
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Placebo | Volanesorsen
Number analyzed (Participants) | 31 | 30
participants | 3 | 23
Statistical Analysis 1: Comparison: Placebo vs Volanesorsen; Test type: Superiority; p = 0.0001, Regression, Logistic; Odds Ratio (OR) = 186.16, 95% CI 2-sided [lower limit 12.86] (NA indicates that the upper limit of 95% CI was not estimable. The upper limit of the odds ratio estimate from the logistic regression model was >999.999, and it was reported as NA per statistical reporting convention.)

5. Secondary Outcome: Treatment Response Rate Defined as Participants With Fasting TG ≥ 40% Reduction From Baseline at Month 3
Description: The Month 3 endpoint was defined as the average of Week 12 (Day 78) and Week 13 (Day 85) fasting assessments.
Time Frame: Baseline to 3 months
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Placebo | Volanesorsen
Number analyzed (Participants) | 33 | 33
participants | 3 | 29
Statistical Analysis 1: Comparison: Placebo vs Volanesorsen; Test type: Superiority; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 99.69, 95% CI 2-sided [15.75 to 631.06]

6. Secondary Outcome: Frequency and Severity of Participant-reported Abdominal Pain During the Treatment Period
Description: Abdominal pain was measured according to the Bracket electronic patient-reported outcomes (ePRO) assessment. Scores were categorized as follows: no pain (pain score: 0), mild (pain score: 1-3), moderate (pain score: 4-6), or severe (pain score: 7-10). The yearly frequency was calculated as the number of episodes during the on-treatment period / (last dose date - first dose date + 28) * 365.25. Missing data were imputed by using next observation carried back (NOCB) if there was a subsequent score available.
Time Frame: Baseline to 12 months
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Placebo | Volanesorsen
Number analyzed (Participants) | 33 | 33
participants
  No pain | 19 | 18
  Mild | 1 | 4
  Moderate | 5 | 6
  Severe | 8 | 5

7. Secondary Outcome: Frequency of the Composite of Episodes of Acute Pancreatitis and Participant-reported Moderate/Severe Abdominal Pain During the Treatment Period
Description: Moderate/severe abdominal pain was defined as having a pain score of 4-10 on the Bracket electronic patient-reported outcomes (ePRO) assessment. Scores were categorized as follows: no pain (pain score: 0), mild (pain score: 1-3), moderate (pain score: 4-6), or severe (pain score: 7-10). The yearly frequency was calculated as the number of episodes during the on-treatment period / (last dose date - first dose date + 28) * 365.25.
Time Frame: 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: events per participant per year
Arm/Group | Placebo | Volanesorsen
Number analyzed (Participants) | 33 | 33
events per participant per year | 2.04 (4.28) | 2.73 (6.57)
Statistical Analysis 1: Comparison: Placebo vs Volanesorsen; Test type: Superiority; p = 0.6131, t-test, 2 sided

8. Secondary Outcome: Change From Baseline in Hepatosplenomegaly as Assessed by MRI at Week 52
Description: The Week 52 endpoint was defined as the average of Week 50 (Day 344)/Week 51 (Day 351) and Week 52 (Day 358) fasting assessments.
Time Frame: Baseline to Week 52
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: cubic centimeters (cm^3)
Arm/Group | Placebo | Volanesorsen
Number analyzed (Participants) | 33 | 33
cubic centimeters (cm^3) | -25 [-150 to 100] | 113 [-43 to 269]
Statistical Analysis 1: Comparison: Placebo vs Volanesorsen; Test type: Superiority; p = 0.1206, ANCOVA; Least Squares Mean Difference = 138, 95% CI 2-sided [-36 to 312]

ADVERSE EVENTS:
Time Frame: Up to approximately 65 weeks.
Description: The safety set included all randomized participants who received at least one dose of study drug.
Arm/Group | Placebo | Volanesorsen
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/33
Serious Adverse Events (participants affected / at risk) | 5/33 | 7/33
Other Adverse Events (participants affected / at risk) | 27/33 | 32/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=33) | Volanesorsen (N=33)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Colitis ischaemic (Gastrointestinal disorders) | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 2 | 0
Cyst (General disorders) | 0 | 1
Cholangitis (Hepatobiliary disorders) | 0 | 1
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Liver function test abnormal (Investigations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=33) | Volanesorsen (N=33)
Injection site erythema (General disorders) | 1 | 25
Injection site pain (General disorders) | 3 | 15
Fatigue (General disorders) | 3 | 7
Injection site swelling (General disorders) | 2 | 7
Asthenia (General disorders) | 3 | 5
Injection site pruritus (General disorders) | 0 | 8
Injection site discolouration (General disorders) | 0 | 7
Injection site induration (General disorders) | 0 | 7
Injection site bruising (General disorders) | 0 | 5
Injection site oedema (General disorders) | 0 | 5
Injection site reaction (General disorders) | 0 | 4
Chest pain (General disorders) | 2 | 1
Influenza like illness (General disorders) | 0 | 3
Injection site hypoaesthesia (General disorders) | 0 | 3
Injection site pallor (General disorders) | 0 | 3
Injection site warmth (General disorders) | 0 | 3
Oedema (General disorders) | 1 | 2
Chills (General disorders) | 0 | 2
Injection site dryness (General disorders) | 0 | 2
Injection site haematoma (General disorders) | 0 | 2
Injection site urticaria (General disorders) | 0 | 2
Malaise (General disorders) | 0 | 2
Pain (General disorders) | 2 | 0
Nasopharyngitis (Infections and infestations) | 7 | 5
Urinary tract infection (Infections and infestations) | 3 | 2
Gastroenteritis (Infections and infestations) | 3 | 1
Influenza (Infections and infestations) | 3 | 1
Bronchitis (Infections and infestations) | 2 | 1
Sinusitis (Infections and infestations) | 1 | 2
Upper respiratory tract infection (Infections and infestations) | 2 | 1
Viral infection (Infections and infestations) | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 6 | 9
Nausea (Gastrointestinal disorders) | 2 | 6
Vomiting (Gastrointestinal disorders) | 3 | 5
Diarrhoea (Gastrointestinal disorders) | 2 | 5
Abdominal pain upper (Gastrointestinal disorders) | 4 | 2
Constipation (Gastrointestinal disorders) | 0 | 2
Flatulence (Gastrointestinal disorders) | 2 | 0
Erythema (Skin and subcutaneous tissue disorders) | 3 | 6
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 3
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 4
Rash (Skin and subcutaneous tissue disorders) | 1 | 3
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 3
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 4
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Headache (Nervous system disorders) | 5 | 7
Hypoaesthesia (Nervous system disorders) | 1 | 2
Paraesthesia (Nervous system disorders) | 0 | 2
Somnolence (Nervous system disorders) | 0 | 2
Platelet count decreased (Investigations) | 1 | 11
Haemoglobin decreased (Investigations) | 2 | 1
Creatinine renal clearance decreased (Investigations) | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 5
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Hypertension (Vascular disorders) | 0 | 3
Hot flush (Vascular disorders) | 2 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 3
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes